CLINICAL TRIAL: NCT04262102
Title: A Quasi-experimental Approach to Characterize the Factors That Influence the Acceptance of New Foods by Infants: Mothers' Diet and Weaning Method: The Dastatuz Project
Brief Title: The Dastatuz Project
Acronym: Dastatuz
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Collaborators: Basque Government Department of Public Health (Other); Bioaraba Health Research Institute (Network); Biodonostia Health Research Institute (Unknown); Biobizkaia Health Research Institute (Other Government)
Responsible Party: Principal Investigator, Olaia Martinez Gonzalez, Associate Professor at the Department of Pharmacy and Food Science of the Faculty of Pharmacy at the University of the Basque Country (Universidad del País Vasco, EHU/UPV)., University of the Basque Country (UPV/EHU)
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: DAST2019
Record Dates: First submitted 2020-01-17; First posted 2020-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Food Preferences; Food Habits; Food Selection
Keywords: Children food neophobia; Fruit and vegetables; Mother's diet; Breastfeeding; Baby-led weaning; Spoon feeding; Nutrition; Weaning
MeSH Terms: conditions — Food Preferences; Feeding Behavior; Breast Feeding

STUDY DESIGN:
Intervention Model Description: After completing the first questionnaire, researchers will allocate each participant into one of the groups (standard diet or high fruit and vegetable diet) depending on their eating habits. Then, when participants' children start with the complementary feeding (spoon-fed or baby-led) chosen by their parents, two new groups will be created. Participants will be allocated to those two new groups depending on the complementary feeding style they have chosen for their children. Therefore, the study will follow the factorial model, created by the following groups: standard diet and spoon-feeding (group 1), standard diet and baby-led weaning (group 2), high fruit and vegetable diet and spoon-feeding (group 3), and high fruit and vegetable diet and baby-led weaning (group 4).
Who Masked: Participant
Masking Description: Single blinding. Participants will not know in which dietary group they belong to (Standard diet or High fruit and vegetable diet). We will give them dietary advice depending on their eating habits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (SD_SF) (Active Comparator): Women will follow a personalized standard diet, described in National Diet Surveys. And their children will be spoon-fed during complementary feeding.
  Interventions: Behavioral: SD_SF
- Group 2 (SD_BLW) (Experimental): Women will follow a personalized standard diet, described in National Diet Surveys. And their children will follow a baby-led weaning approach for complementary feeding.
  Interventions: Behavioral: SD_BLW
- Group 3 (HFV_SF) (Experimental): Women will follow personalized diet, high in fruits and vegetables. And their children will be spoon-fed during complementary feeding.
  Interventions: Behavioral: HFV_SF
- Group 4 (HFV_BLW) (Experimental): Women will follow personalized diet, high in fruits and vegetables. And their children will follow a baby-led weaning approach for complementary feeding.
  Interventions: Behavioral: HFV_BLW

INTERVENTIONS:
Behavioral: SD_SF — Women will follow a personalized standard diet, described in National Diet Surveys. And their children will be spoon-fed during complementary feeding.
  Arms: Group 1 (SD_SF)
Behavioral: SD_BLW — Women will follow a personalized standard diet, described in National Diet Surveys. And their children will follow a baby-led weaning approach for complementary feeding.
  Arms: Group 2 (SD_BLW)
Behavioral: HFV_SF — Women will follow personalized diet, high in fruits and vegetables. And their children will be spoon-fed during complementary feeding.
  Arms: Group 3 (HFV_SF)
Behavioral: HFV_BLW — Women will follow personalized diet, high in fruits and vegetables. And their children will follow a baby-led weaning approach for complementary feeding.
  Arms: Group 4 (HFV_BLW)

SUMMARY:
Unhealthy eating habits are a social challenge in this century, regarding that children usually refuse to eat and taste fruits and vegetables. The Dastatuz project aims to study children food neophobia (the term used referring the reluctance to taste new foods) and fruit and vegetables acceptance. It pretends to tackle the issue from an early stage: pregnancy, lactation and complementary feeding. In this sense, the Project aspires to assess the possible impact of maternal diet and complementary feeding on young children eating behaviour until 18 months of age. In addition, it intends to study the effect that the type of complementary feeding (spoon-fed or baby-led) might have on that eating behaviour. Considering these objectives, a quasi-experimental, multicenter, controlled and prospective intervention study is proposed. If it proved to be effective, this experience would have a high potential to be transferred and would open the possibility to give way to future public programs or guidelines, as a basic and easy solution to achieve higher fruit and vegetable intake among children and, consequently, the potential health benefits this may bring.

Besides, taking into consideration the above mentioned ideas, the investigators hypothesized that a high intake and variety of fruit and vegetables (FV) during pregnancy and breastfeeding will lead to distinctive sensorial experiences for the baby, different from those of the babies whose mothers following a "standard diet" (as described in the National Nutrition Surveys). This consumption profile will promote the acceptance of fruits and vegetables along complementary feeding. Additionally, a correct baby-led weaning (BLW) may also contribute to establish these healthy eating habits.

DETAILED DESCRIPTION:
A quasi-experimental, multicentre, controlled and prospective intervention study is proposed. Guidelines from the TREND (Transparent Reporting of Evaluations with Nonrandomized Designs) statement for non-randomised control trials on behavioural and public health interventions will be followed meticulously in order to follow a realistic scenario which could be easily reproduced onwards. Initially, mothers in the third trimester of pregnancy (n=384) will be assigned to different diet profiles according to their own food preferences (Standard diet, SD vs. High Fruit and Vegetable diet, HFV); next, caregivers' willingness to perform weaning following one or other approach will be the base to establish groups (Spoon feeding, SF vs. Baby Led Weaning, BLW, respectively). Regardless of their distribution, all of them will receive the current standard recommendations and care. Intervention groups will receive additional diet recommendations during pregnancy, breastfeeding and weaning. The study implies a time period from the third trimester of the pregnancy until children are 18 months old. Follow-up, sampling and/or measurements will be performed at 6-7th months of pregnancy, before delivery; 2nd, 4th, 6th, 12th and 18t months from birth. Moreover, 5-6 meetings are going to be held either at the Outpatient Consultation of the Txagorritxu Hospital (Vitoria-Gasteiz) or at the Faculty of Psychology of the University of the Basque Country (Donostia-San Sebastian), where material and information are going to be given to the participants.

Procedure Baseline questionnaire and dietary assessment will be the base for group blind assignment. Those below the national (Spain) mean consumption of fruits and vegetable (about 414 g/person/day) or/and those who claim to have difficulties achieving the recommended portions will be included in the control group (SD, see arms of the intervention). When a fruit consumption of one standard deviation bellow the mean is detected, dietetic assessment will be performed in order to encourage, at least, the mean intake. Those above the national (Spain) mean consumption of fruits and vegetable (about 414 g/person/day) will be included in the experimental group (HFV, see arms of the intervention). During the study, they will be encouraged and assessed to achieve even a higher intake, 800 g/person/day. If a significant FV decrease in their diet is detected in the follow-ups, dietetic assessment will be performed in order to restore the initial intake. For weaning groups, those better disposed to follow a spoon-feeding approach will be included in the control group (SF, see arms of the intervention); and those better disposed to follow a baby-led approach will be included in the intervention group (BLW, see arms of the intervention).

Several measuring tools are proposed to obtain objective data along the designed project:

QUESTIONNAIRES

* Q1: Participants will complete this questionnaire during recruitment and it will collect information about their socio-economic and psychological status, her actual diet profile and her expectations about the feeding of her future baby. It will also contain a question regarding preferred contact method (email/telephone/post).
* Q2: This is a follow-up questionnaire (completed by online questionnaires) which will assess the adherence to the diet of the mother along pregnancy. Moreover, it will also collect information about the psychological aspect, such as the parental stress level of participants.
* q1: It is a short questionnaire on the breastfeeding efficacy that will be completed on the second week post-partum. It has been used to predict breastfeeding duration and exclusivity.
* Q3: It is very similar to the Q2 questionnaire, but parameters will be studied during lactation.
* Q4: This will also be a follow-up questionnaire. Although it is quite similar to Q3, this one includes a new questionnaire about parental feeding styles.

SAMPLES: Milk samples from the mothers will be collected along the second or third month of breastfeeding. Instructions will be given to the mothers as follows: collect approximately 50mL-100mL in a sterilized container and freeze it (-20ºC) within 5 min of expression; if the samples are going to be delivered right after the extraction they could be maintained at 4ºC. Participants will be given sample carrier and transporting containers in order to deliver them to one of the two collection points of the Biobanco. Samples will be transported to the main center of the Biobanco in Galdakao and maintained frozen at -25ºC until analysis in which composition profile and viscosity and other physical properties (i.e. shear stress) will be assessed by Infrared Spectroscopy MilkoScan (Foss Electric, Denmark), gas chromatographic- mass spectrometry (GC-MS) and rheometry techniques (rheometer AR1000, TA Instruments). Nutritional analysis will be carried out at the Galdakao center of the Biobanco and rheological analysis at the Faculty of Pharmacy of the Unviersity of the Basque Country.

OBSERVATIONS: At 6, 8 and 12 months from birth, prior to paediatric consultation, each family will record for 24h the food intake of the child indicating: food consumed and its composition or commercial brand, if necessary; family will also report cooking method and will record the weight of food consumed.

Some days after the paediatric control of the 6th, 8th and 12th month parents will be contacted by phone to gather information about foods which might be new for the child, and therefore, has never tried them. According to the answers received, some recipes will be sent by e-mail to each family, together with instructions of how to offer these foods to the baby (moments, times, circumstances). Parents will be asked to record a video of these mealtimes and send to the research team. Times swallowed and acceptance or rejection signs will be studied. These records will only be used for research purposes stated in this project, and always previous informed consent signed by the parents or tutors of the child. In addition, Q4 will be sent to the families, by email, as an online questionnaire. It will gather information from the parents about the eating behaviour of the child. This last questionnaire will also record weight/height data and psychological features of the child.

ALLERGEN RISK: In addition to the above mentioned measurements, allergen risk will be assessed comparatively (spoon diet vs baby led), following general risk assessment procedures. This is a well characterized gap which remains understudied, as it is recognised in the literature. Exposition analysis will be performed using data from the 24 hours diet records until 12 months from birth. Main allergens, mentioned at Regulation 1169/2011 (CE) of the European Parliament and of the Council of 25 October 2011on the provision of food information to consumers, will be assessed. Moreover, especial attention will be paid to FODMAPS, which today arise interest as a potential reason to the permanence of celiac-like symptoms, even when in theory a gluten free diet is being correctly followed. Analysis will be based on the 24h food diary transmitted by families. Ingredients used on the meals preparation will be taken into consideration. A procedure established by the Food Standard Agency will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy mothers who are notified about the study (and express interest to take part) before week 24 of gestation.
* Spanish, Basque or English speakers.
* Intention to live in the Basque Country until the child will be 18 months old.
* Age: 18-45 years.

Exclusion Criteria:

* Unhealthy mother or complicated pregnancy (all types of diabetes mellitus, high blood pressure, etc.).
* Not willing to breastfeed.
* Mother with too much diet restrictions and detection of severe non-adherence to the diet prescribed and any condition contraindicated for the development of the project.

After birth, women will be excluded if:

* Their infant is born before 37 weeks gestation
* Their infant is born with a congenital abnormality, physical condition, or intellectual disability, which was likely to affect the infant's feeding or growth is identified.

Also, there will not be any milk collection from mothers who are taking any medication.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 384 (Estimated)
Dates: Start 2019-10-18 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Change of diet during pregnancy and breastfeeding: predimed | Baseline, 8-9th month of pregnancy, 4th month after delivery, 6th month after delivery
  This possible change will be measured using Predimed questionnaire (Martínez-González et al., 2012), which has 14 items that evaluate adherence to the Mediterranean Diet. Each of the items has a different criterion to get a point, being 0 the minimum and 14 maximum of the total score. If total score is ≤7, it means low adherence; if total score is >7, it means high adherence.
Change of diet during pregnancy and breastfeeding: precoded food record | Baseline, 8-9th month of pregnancy, 4th month after delivery, 6th month after delivery
  This possible change will be measured using Pre-coded Food Record Form (Rodriguez et al., 2014), which gives information about the intake of foods in portions per day.
Change of fruit and vegetable intake | Beginning of the weaning process (it will depend upon each participant, from 4th month to 6th month), 6th month after delivery, 12th month after delivery, 18th month after delivery
  Measured by an ad hoc questionnaire reported by parents.
Change of food acceptance of exposed fruits and vegetables as the measurement of willingness to eat them | 6th month after delivery, 12th month after delivery, 18th month after delivery
  Assessed by videotaped meals of children.

SECONDARY OUTCOMES:
Composition profile of mother´s milks (1) | 2nd month after delivery
  Measured by Infrared Spectroscopy MilkoScan (Foss Electric, Denmark) to measure nutritional composition of the milk samples (mg nutrient/100 mL).
Composition profile of mother´s milks (2) | 2nd month after delivery
  Measured by Gas chromatographic- mass spectrometry (GC-MS) to measure aromatic profile of the milk samples (ppm).
Rheological characteristics of mother´s milks | 2nd month after delivery
  Measured by Rheometry techniques (rheometer AR1000, TA Instruments) to measure apparent viscosity in (mPa•s).
Child´s diet profile | Beginning of the weaning process (it will depend upon each participant, from 4th month to 6th month), 6th month after delivery, 12th month after delivery, 18th month after delivery
  Measured by 24h dietary recall reported by parents.
Child´s nutritional state | Beginning of the weaning process (it will depend upon each participant, from 4th month to 6th month), 6th month after delivery, 12th month after delivery, 18th month after delivery
  Assessed by the periodical paediatric control, reported then by parents.
Adherence to the diet assigned to each group | 8-9th month of pregnancy, 4th month after delivery
  Measured by Pre-coded Food Record Form (Rodriguez et al., 2014).
Children BMI from birth | 6th, 9th and 12th months after birth, following the paediatric callendar.
  Assessed by the periodical paediatric control, reported then by parents.
Mother's psychological state regarding pregnancy | Baseline
  Assessed by Prenatal Evaluation Questionnaire (Armengol Asenjo et al., 2007), composed by 42 items divided in 7 dimensions: (1) pregnancy acceptance, (2) identification of the maternal role, (3) quality of the relationship with her mother, (4) quality of the relationship with her partner, (5) preparation for labour, (6) fear to pain and loss of control during labour, and (7) preoccupation for her and her baby's wellbeing. Possible answers are: A=a lot, B= with frequency, C= sometimes, and D= never (Likert scale, from 1 to 4 points).
Maternal anxiety | Baseline, 8th-9th month of pregnancy, 4th month after delivery, 6th month after delivery
  Assessed by State-Trait Anxiety Inventory (STAI) questionnaire (Jover et al., 2014). It is composed by 20 items and answers are given on a 4-point Likert scale (0= absolutely not and 4= very much). A high score indicates a higher anxiety.
Level of depression | Baseline, 8th-9th month of pregnancy, 4th month after delivery, 6th month after delivery
  Assessed by the Edinburgh Postnatal Depression Scale (EDPS) (Garcia-Esteve et al., 2003). This questionnaire composed by 10 items (answered punctuated 0-3 depending on symptoms severity) will show us the level of depressive symptoms participants present.
Breastfeeding efficacy and certainty | Week 2 after delivery, 4th month after delivery
  Assessed by the Breastfeeding Self-Efficacy Scale (Oliver-Roig et al., 2012). Punctuation is set in a 5-point Likert-type scale where 1 indicates not at all confident and 5 indicates always confident. The higher the score, the higher level of breast- feeding self-efficacy.
Parental feeding styles | 6th month after delivery, 12th month after delivery, 18th month after delivery
  Assessed by the Parental Feeding Styles questionnaire (Wardle et al., 2002). 27 items are divided in four subscales: emotional feeding, instrumental feeding, encouragement to eat new foods, and control over eating. Answer range goes from 1= never to 5= always. A high score in each subscale means a higher level on that issue.
Acceptance of novel foods (1) | 6th month after delivery, 12th month after delivery, 18th month after delivery
  Assessed by an ad hoc questionnaire.
Acceptance of novel foods (2) | 6th month after delivery, 12th month after delivery, 18th month after delivery
  Assessed by videotaped meals. The Feeding Infants: Behaviour and Facial Expression Coding System (FIBFECS) (Hetherington et al., 2016) will be taken into consideration for this issue.

CONTACTS AND LOCATIONS:
Overall Officials: Olaia Martinez Gonzalez, PhD, Principal Investigator — University of the Basque Country/ Basque Country University; Edurne Maiz Aldalur, PhD, Principal Investigator — University of the Basque Country/ Basque Country University
Locations (2):
- Spain (2):
  - Pharmacy and Food Science Department of the Basque Country/Basque Country University (Universidad del País Vasco, UPV/EHU)., Vitoria-Gasteiz, Spain/Alava
  - and Department of Personality Assessment and Psychological Treatments of the Faculty of Psychology of the University, Donostia / San Sebastian, Spain/Guipuzcoa

REFERENCES:
- [Derived] Urkia-Susin I, Rada-Fernandez de Jauregui D, Orruno E, Maiz E, Martinez O. A quasi-experimental intervention protocol to characterize the factors that influence the acceptance of new foods by infants: mothers' diet and weaning method. Dastatuz project. BMC Public Health. 2021 May 13;21(1):918. doi: 10.1186/s12889-021-10967-7. PMID 33985471